# **STUDY DOCUMENT**

Official Study Title:

The Effect of Prone Position on Oxygen Saturation, Blood Gas Parameters, and Respiratory Rate in Intensive Care Patients with COVID-19-induced ARDS

NCT Number: NCTXXXXXXX

Document Type: Study Protocol

Document Date: 26 May 2025

#### STUDY PROTOCOL

### 1. Oficial Title

The Effect of Prone Position on Oxygen Saturation, Blood Gas Parameters, and Respiratory Rate in Intensive Care Patients with COVID-19-induced ARDS

#### 2. Brief Title

Effect of Prone Position in COVID-19 ARDS Patients

## 3. Principal Investigator(s)

- Dr. Veysel Tekin, RN, Ph.D. Diyarbakır Provincial Health Directorate
- Prof. Dr. Medet Korkmaz, RN, Ph.D. Inonu University Faculty of Nursing

## 4. Study Sites

General and Intermediate Intensive Care Units, Eastern Turkey

## 5. Study Period

Start Date: April 1, 2021 End Date: August 30, 2021

# 6. Background and Rationale

ARDS is a common complication of severe COVID-19, associated with high mortality. Prone positioning has been shown to improve oxygenation and lung compliance in ARDS. This study investigates its short-term effectiveness in non-intubated patients.

### 7. Objectives

To evaluate the impact of a 30-minute prone position on:

- Oxygen saturation (SpO<sub>2</sub>, SaO<sub>2</sub>, PO<sub>2</sub>)
- Respiratory rate
- Blood gas parameters (pH, PCO<sub>2</sub>, Lactate, Sodium)

### 8. Study Design

Randomized controlled trial

Parallel group, repeated measures (6 total timepoints)

1:1 allocation (n = 90, 45 per group)

#### 9. Eligibility Criteria

- \*\*Inclusion Criteria:\*\*
- Age ≥ 40
- ICU hospitalization for COVID-19-induced ARDS
- Intubated and responsive to assessment
- \*\*Exclusion Criteria:\*\*
- Sensory impairments (vision/hearing)

- Cognitive impairments
- Patients who died or no longer required ICU during study

#### **10.** Intervention

- \*\*Experimental Group:\*\* 30 minutes prone position once daily for 2 days
- \*\*Control Group:\*\* Supine standard care

#### 11. Outcomes

- \*\*Primary Outcome:\*\*
- Change in oxygen saturation (SpO<sub>2</sub>) post-prone positioning
- \*\*Secondary Outcomes:\*\*
- Respiratory rate
- Arterial blood gas values (SaO<sub>2</sub>, PO<sub>2</sub>, PCO<sub>2</sub>, pH, lactate, sodium)

#### 12. Randomization

Simple randomization by drawing lots

Allocation ratio 1:1

### 13. Blinding

Open-label (no blinding)

#### **14. Statistical Methods**

Paired and independent t-tests Wilk's Lambda Cohen's d for effect size SPSS used for data analysis

### **15. Ethical Considerations**

Approval: Gazi Yasargil Training and Research Hospital Ethics Committee (15.01.2021 / No: 626)

Verbal and written consent obtained Conducted per Declaration of Helsinki

# **16. Data Sharing Plan**

Available upon reasonable request from the corresponding author.